CLINICAL TRIAL: NCT03955991
Title: Stress Management Effects on Affective Status and Influenza Vaccine Response in Older Breast Cancer Patients
Brief Title: VSMART (Video-Conference Stress Management and Relaxation Training for Older Women With Breast Cancer)
Acronym: VSMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Principal Investigator, Michael H. Antoni, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160525
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-06

CONDITIONS: Stress
Keywords: Breast Cancer; Flu Vaccine
MeSH Terms: conditions — Breast Neoplasms; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- R-CBSM (Experimental): 10 weeks of group intervention convene by a broadband connection for approximately 75-90 minutes. Intervention given prior to Influenza Vaccine.
  Interventions: Behavioral: R-CBSM; Biological: Influenza vaccine
- Wait List Condition (WLC) (Active Comparator): Persons assigned to this group will receive R-CBSM approximately 28 days after receiving the Influenza Vaccine.
  Interventions: Behavioral: R-CBSM; Biological: Influenza vaccine

INTERVENTIONS:
Behavioral: R-CBSM — 10 weekly educational modules via an electronic tablet. A participant workbook is also provided that contains a summary of the rationale for each module, outline of each technique, and homework exercises.
Biological: Influenza vaccine — Standard of care Influenza vaccine for that given year.

SUMMARY:
The proposed study tests the effects of a novel remotely-delivered group cognitive behavioral stress management (R-CBSM) intervention on improving health and quality of life in older women undergoing breast cancer (BCa) treatment. This study tests if delivered home-based group CBSM (R-CBSM) improves response to influenza vaccine (IV) in parallel with improved psychological adaptation, inflammation and other immune functioning indicators in older women treated for BCa.

ELIGIBILITY:
Inclusion Criteria:

1. Must meet the criterion of a score of >14 on the Impact of Event Scale-Intrusion scale (IES-I48) for cancer-specific distress or self-report at least moderate distress (score of 4 or greater) on a screening question, "How would you rate your distress level, over the past week, on a scale of 0 to 10, with 0 meaning no distress and 10 being extreme distress"
2. No prior history of cancer (with the exception of non-melanoma skin cancer)
3. Life expectancy of > 12 months.
4. No diagnosis of major psychiatric condition or mental disorder (i.e. schizophrenia, psychosis, and/or bipolar disorder) or active (in the past 12 months) Major Depressive Disorder (MDD), panic disorder, Post Traumatic Stress Disorder (PTSD) diagnosis or history of suicide thoughts, attempts or plans.
5. No substance dependency in the past 12 months.
6. No acute or chronic co-morbid medical condition with known effects on the immune system (e.g., HIV infection, autoimmune diseases)
7. No prior neo-adjuvant therapy
8. No current medications that act as direct immunomodulators (e.g., Granulocyte Macrophage Colony Stimulating Factor (GM-CSF), interferons)
9. No significant cognitive impairment, must score <31 on the Telephone Interview for Cognitive Status (TICS)49.
10. At least a 6th grade reading level in English and be available for follow-up
11. Women age 50 and older diagnosed with stage 0-III breast cancer.

Exclusion Criteria:

* Does not meet all Inclusion Criteria.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Hemagglutination inhibition assay (HAI) - Fold response to IV | 28 days post vaccine
  As measure HAI antibody titers change from pre-vaccine to 28 days post vaccine
Percent of cases that achieve a clinical vaccine response of greater than or equal to 4 fold titer increase. | 28 days post vaccine
  Participant's score will be dichotomized into whether 4 fold increase was achieved. Via serum.

SECONDARY OUTCOMES:
Change in Affective Status | Baseline (T0), 6 months (T1), 7-days post IV (T2), 28-day post IV (T3), 12 month post Baseline (T4).
  Affective Status is comprised of the Impact of Event Score Intrusion (IES-I), Affect Balance Scale (ABS) negative affect, positive affect and Center for Epidemiologic Studies Depression (CES-D) that comprise a latent construct
Change in Circulating Cytokine levels | Baseline (T0), 6 months (T1), 7-days post IV (T2), 28-day post IV (T3)
  Serum from blood samples will be evaluated for cytokine indices for Interleukin
  (IL) 1, IL-6 and Tumor Necrosis Factor (TNF-Alpha).
Change in Affective Status markers | Baseline (T0) to 28-day post IV (T3).
  Affective status change as measured by a Latent variable that compares the effects of the 2 groups.
Change in Immune Status measured by Activation Induced Cytidine Deaminase (AID) in response to Cytosine-phosphate -Guanine (CpG) | Baseline (T0) to 6 months (T1).
  Level of AID activity in B cells
Change in Immune Status measured by Switched B-cells (swB) | Baseline (T0) to 28-day post IV (T3).
  Percentage of B-cells indicator.
Magnitude of Immune changes associated with Flu Vaccine response | Baseline (T0) to 28-day post IV (T3)
  Measured by a change score in sw B-Cell and AID response with change HAI response
Magnitude of Inflammatory changes associated with Flu Vaccine response | Baseline (T0) to 28-day post IV (T3)
  Measured by a change score in inflammatory cytokines with change in HAI response

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Antoni, Ph.D, Principal Investigator — University of Miami
Locations (1):
- Flipse Building, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saez-Clarke E, Walsh EA, Lovan P, Plotke R, Ream M, Popok P, Perdomo D, Blomberg B, Antoni MH. Distress tolerance and perceived cancer-related cognitive impairment in nonmetastatic breast cancer. Health Psychol. 2025 Feb;44(2):166-170. doi: 10.1037/hea0001417. Epub 2024 Sep 23. PMID 39311813